CLINICAL TRIAL: NCT07071961
Title: Regorafenib (Reg) and Lorigerlimab (Lor), RELO Regimen, in Treatment of High-risk Patients With Colorectal Cancer With Radiographic Occult Molecular Residual Disease After End of Established Definitive Therapy [ReLOAD Trial]
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bayer (Industry); MacroGenics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1853; NCI-2025-05156 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2025-07-16; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Cancer; Regorafenib; High Risk Patients
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- RELO in ctDNA+ mCRC (Experimental): receive regorafenib and lorigerlimab for up to 6 months
  Interventions: Drug: Regorafenib (CT); Drug: Lorigerlimab

INTERVENTIONS:
Drug: Regorafenib (CT) — Given by po
Drug: Lorigerlimab — Given by IV

SUMMARY:
To learn about the effects of the drugs regorafenib and lorigerlimab on circulating tumor DNA (ctDNA) in patients with CRC and who have radiographic occult minimal residual disease (MRD) after completing standard-of-care therapy

DETAILED DESCRIPTION:
Primary Objectives

• To determine the 6-month circulating tumor (ctDNA) clearance rate following 6 months of therapy with RELO regimen in patients with colorectal cancer (CRC) who present with radiographic occult molecular residual disease (MRD) after completing definitive standard-of-care (SOC) therapy.

Secondary Objectives

* To determine the 3-month ctDNA clearance rate following RELO treatment.
* To determine disease-free survival (DFS) following 6 months of RELO treatment.
* To determine overall survival (OS) following 6 months of RELO treatment.
* To determine the safety and tolerability of RELO.

ELIGIBILITY:
Eligibility Criteria

* Histological confirmation of CRC
* Post-R0 resection of stages II, III, or IV CRC and all planned adjuvant therapies have been completed.
* No evidence of radiographic disease within 28 days (before or after) of a positive ctDNA assay
* Evident MRD as defined by positive ctDNA assay. Participants may be identified for enrollment with any Clinical Laboratory Improvement Amendments (CLIA)-certified ctDNA assay for MRD. MRD status will be confirmed with the Signatera assay prior to initiation of therapy (unless the prior testing was also done with Signatera in which case this test would not require confirmation)
* Adequate organ and marrow function as defined below:

  * Absolute neutrophil count: ≥1,000/mcL
  * Platelets: ≥100,000/mcL
  * Total bilirubin ≤1.5 x the upper limit of normal (ULN). Total bilirubin (≤3 x ULN) is allowed if Gilbert's syndrome is documented.
  * AST(SGOT)/ALT(SGPT): ≤3 × institutional ULN (≤5 x ULN for participants with liver involvement of their cancer).
  * Creatinine clearance ≥40 mL/min. Creatinine clearance (Clcr) can either be measured in a 24-hour urine collection or estimated by the Cockcroft-Gault equation as follows: Clcr (mL/min) = [(140 - age) x (weight in kg) ÷ [72 x (serum creatinine in mg/dL)] [0.85 if female]
* ECOG performance status (PS) of 0 or 1
* Age ≥ 18 years. Because no dosing or adverse event data are currently available on the use of regorafenib in these participants, children <18 years of age are excluded from this study.
* Able to understand and is willing to sign a written informed consent document.
* The effects of RELO on the developing human fetus are unknown. For this reason and because regorafenib appears to be teratogenic in animal models, women of child-bearing potential (refer to MDA Policy CLN 1114) must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry, for the duration of study participation and for at least 4 months after the last dose. This includes all female participants, between the onset of menses (as early as 8 years of age) and 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following:

O Postmenopausal (no menses in greater than or equal to 12 consecutives months).

* History of hysterectomy or bilateral salpingo-oophorectomy.
* Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal
* range, who have received Whole Pelvic Radiation Therapy).
* History of bilateral tubal ligation or another surgical sterilization procedure.) Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice, however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of administration

Exclusion Criteria

* Concurrent treatment with drug with which the interactions are considered clinically significant by investigator (as outlined in section 0). Major surgical procedure or significant traumatic injury within 21 days before start of study medication. Note: If participants received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Grade 2 or higher peripheral neuropathy per CTCAE v5.0.
* Systemic therapy with immunosuppressive agents within 7 days or use of any investigational drug within 28 days before the start of trial treatment except for participants who may be receiving low dose prednisone (specifically receiving ≤10 mg prednisone or equivalent within 7 days of treatment initiation).
* Prior exposure to any immune checkpoint blockade agent or any other immunomodulatory agent used for antineoplastic therapy for mCRC.
* Previous malignant disease (other than the target malignancy to be investigated in this trial) within 3 years prior to study treatment initiation.
* Receipt of any organ transplantation, including allogeneic stem cell transplantation (exception: transplants that do not require immunosuppression, such as hair transplant).
* Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent. The study will allow replacement therapy with thyroxine, insulin or physiologic corticosteroid replacement therapy for autoimmune conditions that are well-controlled.
* Known severe hypersensitivity reactions to monoclonal antibodies (Grade ≥ 3 NCICTCAE v5.0), any history of anaphylaxis, or recent (within 5 months) history of uncontrolled asthma.
* Clinically significant cardiovascular/cerebrovascular disease as follows: cerebral vascular accident/stroke (<6 months prior to enrollment), myocardial infarction (<6 months prior to enrollment), unstable angina, congestive heart failure (New York Heart Association Classification Class >II), myocarditis, or serious cardiac arrhythmia.
* Clinically relevant diseases (for example, inflammatory bowel disease) and / or uncontrolled medical conditions, which, in the opinion of the Investigator, might impair the subject's tolerance or ability to participate in the trial.
* Failure to recover from any other toxicity (other than immune-related toxicity) related to previous anticancer treatment to ≤ Grade 2 per CTCAE v5.0.
* Receipt of a live-virus vaccine within 30 days prior to first dose of study drug (seasonal flu vaccines that do not contain live virus are permitted). Patient should refrain to receive live-virus vaccines for 120 days following the last dose of lorigerlimab.
* Evidence of any serious bacterial, viral (active HIV, HCV or HBV), parasitic, or systemic fungal infections within the 30 days prior to the first dose of study drug.
* Subject is pregnant or breast feeding or planning to become pregnant while enrolled in the study, up to the final EOT visit.
* History of (non-infectious) pneumonitis that required steroids, ongoing pneumonitis, or history of interstitial lung disease.
* History of GI perforation or GI bleeding within 4 weeks, significant diverticulitis or flare within 4 weeks, and acute pancreatitis within 4 weeks.
* Grade > 3 (per CTCAE v5.0) proteinuria (> 3.5 g/24 hours)
* Grade > 3 (per CTCAE v5.0) hypertension (systolic blood pressure > 160 or diastolic blood pressure > 100).
* Evidence or history of bleeding diathesis or coagulopathy within 6 months of start of treatment. Subjects with clinically significant thrombotic, embolic, venous, orarterial events, deep vein thrombosis or pulmonary embolism within 6 months of start of treatment. Participants with incidental findings that have started anticoagulation and are stable are allowed.
* Ongoing infection > Grade 2 NCI-CTCAE v5.0.
* Symptomatic metastatic brain or meningeal tumors.
* Presence of a non-healing wound, non-healing ulcer, or bone fracture.
* Major surgical procedure or significant traumatic injury within 28 days before start of study medication
* Renal failure requiring hemodialysis or peritoneal dialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Kanwal Raghav, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org